CLINICAL TRIAL: NCT05778123
Title: Multiomic Analysis of Body Fluid in Acute Traumatic Brain Injury
Acronym: MOSS-FAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Director of Brain Injury Center, RenJi Hospital
Other Study IDs: LY2023-018-B
Record Dates: First submitted 2023-02-05; First posted 2023-03-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Brain Injuries, Traumatic
Keywords: Traumatic brain injury; Body fluid; Biomarker; Multiomic analysis
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI: Patients with traumatic brain injury.
  Interventions: Other: Type of disease
- Control: Patients with hydrocephalus.
  Interventions: Other: Type of disease

INTERVENTIONS:
Other: Type of disease — Different types of pathogen: brain injury by trauma or hydrocephalus due to various diseases.

SUMMARY:
The goal of this experimental observation study is to figure out differently expressed biomarkers in body fluid in traumatic brain injury patients. The main questions it aims to answer is:

* Which RNA, protein and metabolites are differently expressed in lesion tissues?
* What molecular mechanism is participated in TBI? Participants will be treated by emergency operation, and their body fluid samples will be collected in emergency room and during the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and <65
2. Within 12 hours after brain injury
3. Control group is hydrocephalus
4. GCS ≥3 and ≤8
5. Closed brain injury with frontotemporal contusion
6. Need emergency intracranial hematoma evacuating or cerebrospinal fluid shunting operation
7. Patient's agents are informed and consent the research

Exclusion Criteria:

1. With TBI, stroke, ICH or intracranial tumor history
2. Death within 24 hours
3. Immunosuppression state
4. Severe organ dysfunction
5. Complicated infective disease
6. Pregnant

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe traumatic brain injury or hydrocephalus.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
RNA biomarkers in patients' blood & cerebrospinal fluid assessed by transcriptome bioinformatic analysis | Immediately after collecting blood & cerebrospinal fluid
  Patients' blood and cerebrospinal fluid will be collected in emergency room and operation room respectively. Then these samples will be immediately prepared to be detected through transcriptome sequencing. The results of transcriptome sequencing will be further analyzed and compared with control group to filter potential RNA biomarkers in blood and cerebrospinal fluid of severe TBI patients.
Protein biomarkers in patients' blood & cerebrospinal fluid assessed by proteomic bioinformatic analysis | Immediately after collecting blood & cerebrospinal fluid
  Patients' blood and cerebrospinal fluid will be collected in emergency room and operation room respectively. Then these samples will be immediately prepared to be detected through proteomics mass spectrometry. The results of proteomic will be further analyzed and compared with control group to filter potential protein biomarkers in blood and cerebrospinal fluid of severe TBI patients.
Metabolite biomarkers in patients' blood & cerebrospinal fluid assessed by metabolomic bioinformatic analysis | Immediately after collecting blood & cerebrospinal fluid
  Patients' blood and cerebrospinal fluid will be collected in emergency room and operation room respectively. Then these samples will be immediately prepared to be detected through metabolomic mass spectrometry. The results of metabolomic will be further analyzed and compared with control group to filter potential metabolite biomarkers in blood and cerebrospinal fluid of severe TBI patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Injury Center, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No